CLINICAL TRIAL: NCT07141264
Title: A Single-Arm, Exploratory Study of Adebrelimab Combined With Etoposide Capsules as Maintenance Therapy in Extensive-Stage Small Cell Lung Cancer
Brief Title: Adebrelimab Combine With Etoposide Capsules in ES-SCLC Maintenance Therapy
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Tang-Du Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IIT20250816
Record Dates: First submitted 2025-08-19; First posted 2025-08-26 (Actual); Last update posted 2025-12-30 (Actual); Status verified 2025-12

CONDITIONS: SCLC,Extensive Stage
Keywords: SCLC; Adebrelimab; Etoposide Capsules; Maintenance Therapy
MeSH Terms: interventions — Etoposide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Drug: Adebrelimab combined with Etoposide Capsules — Each treatment cycle spans 3 weeks. Sequential medication administration begins on the first day of each cycle: Adebrelimab is administered at a dosage of 1200mg on day 1, every 3 weeks, while Etoposide Capsules is given orally at a dosage of 50mg or 25mg daily, day 1 to 14 of a 21-day cycle. Administration timing allows for a window of ±5 days. Subjects are required to undergo comprehensive assessments, including vital signs monitoring, anthropometric measurements, physical examinations, laboratory analyses, and performance status evaluations, to assess treatment tolerability for continuation.

SUMMARY:
This prospective clinical study aims to evaluate and observe the efficacy and safety of adebrelimab combined with etoposide capsules in maintenance therapy for extensive-stage small cell lung cancer using a single-arm trial design.

The study is planned to be conducted in Shaanxi Province, China, with an initial target enrollment of 32 patients. The study commenced in August 2025, and recruitment is expected to conclude around December 2026, with the trial anticipated to end by December 2027. Assuming no occurrences such as withdrawal of informed consent by subjects, intolerable adverse drug reactions, or investigator-assessed unsuitability for further participation, each participant's estimated duration of study treatment will continue until radiographically confirmed tumor progression.

ELIGIBILITY:
Inclusion Criteria:

1. Voluntary participation with signed informed consent and good compliance for follow-up.
2. Age between 18 and 75 years old.
3. Histologically or cytologically confirmed extensive-stage small cell lung cancer (ES-SCLC) according to the AJCC 8th edition or VALG phase II staging criteria.
4. ECOG performance status score: 0 to 2.
5. Absence of disease progression after receiving 4-6 cycles of platinum-based chemotherapy combined with Adebrelimab induction therapy.
6. Recovery of non-hematologic adverse reactions to grade 1 (except for alopecia, skin pigment changes, or as determined by the investigator) following induction therapy.
7. Time from the end of induction treatment (last dose) to initiation of maintenance treatment ≤ 6 weeks.
8. At least one measurable lesion assessed by the investigator according to RECIST 1.1.
9. Normal function of major organs, meeting the following criteria:

(1)Bone marrow function: Absolute neutrophil count (ANC) ≥ 1.5×10^9/L (grade 1 according to CTCAE 5.0); platelets ≥ 100×10^9/L; hemoglobin > 80g/L.

(2)Renal function: Creatinine ≤ 1.5 times the upper limit of normal (ULN), grade 1 according to CTCAE. Note: If creatinine is greater than 1.5 times the ULN, creatinine clearance must be > 50ml/min.

(3)Liver function: Bilirubin ≤ 1.5 times ULN (grade 1 according to CTCAE), patients with Gilbert's syndrome bilirubin ≤ 3.0 times ULN; AST and ALT ≤ 3.0×ULN.

(4)Coagulation indicators: International normalized ratio (INR) ≤ 1.55 (if the patient is receiving a stable dose of therapeutic warfarin or low molecular weight heparin, INR is usually between 2 and 3), PTT < 1.2 times ULN.

10.Women of childbearing potential must agree to use contraception during the study and for 6 months after the end of the study (such as an intrauterine device, contraceptive pills, or condoms); serum or urine pregnancy test must be negative within 1 week before enrollment, and must be non-lactating patients; men must agree to use contraception during the study and for 6 months after the end of the study.

Exclusion Criteria:

1. Limited-stage small cell lung cancer (SCLC);
2. Histologically or cytologically confirmed mixed histology SCLC;
3. Prior treatment with anti-angiogenic agents;
4. Conditions that may affect oral drug intake, such as inability to swallow, chronic diarrhea, or intestinal obstruction;
5. Major surgery, open biopsy, or significant traumatic injury within 4 weeks prior to enrollment;
6. Participation in another investigational drug clinical trial within 4 weeks prior to enrollment;
7. Relevant medical history:

(1)Untreated or symptomatic brain metastases or spinal cord compression; (2)Concurrent active malignancy requiring treatment; (3)Active autoimmune disease or immunodeficiency, or a history of such conditions, including but not limited to autoimmune hepatitis, interstitial lung disease, uveitis, rheumatoid arthritis, inflammatory bowel disease, hypophysitis, vasculitis, or nephritis.Exceptions include: patients with stable disease not requiring systemic immunosuppressive therapy, such as type I diabetes mellitus, hypothyroidism controlled with hormone replacement therapy, or skin disorders not requiring systemic treatment (e.g., vitiligo, psoriasis, or alopecia), or those with no external triggering factors and a low risk of recurrence; (4)History of psychiatric or substance abuse disorders that would interfere with study compliance; 8.Presence of any severe and/or uncontrolled comorbid conditions, including but not limited to:

1. Uncontrolled hypertension (systolic BP ≥150 mmHg or diastolic BP ≥100 mmHg);
2. Myocardial ischemia or infarction of grade I or higher, arrhythmias (including QTc ≥450 ms in males, ≥470 ms in females), congestive heart failure of NYHA class ≥2, or left ventricular ejection fraction (LVEF) <50% on echocardiogram;
3. Decompensated diabetes mellitus or other contraindications requiring high-dose corticosteroids;
4. Exacerbation of chronic obstructive pulmonary disease (COPD) or other serious respiratory disorders requiring hospitalization;
5. Active or uncontrolled severe infection (≥CTCAE grade 2);
6. Uncontrolled pleural, pericardial, or peritoneal effusion requiring repeated drainage;
7. Liver cirrhosis, decompensated liver disease, active hepatitis, or chronic hepatitis requiring antiviral treatment;
8. Renal insufficiency: urine protein ≥++ on routine urinalysis and 24-hour urine protein >1.0 g confirmed; 9.Severe infection within 4 weeks before the first dose, including but not limited to infectious complications, bacteremia, severe pneumonia requiring hospitalization, or infections requiring intravenous antibiotics, antifungals, or antivirals; or unexplained fever >38.5°C during screening or prior to first dose; 10.Grade III-IV immune-related adverse events (irAEs) during the induction phase with PD-L1 inhibitors; 11.Active brain or leptomeningeal metastases at enrollment; Exception: patients who received prior treatment (e.g., radiotherapy) for brain or leptomeningeal metastases during or before induction and had stable disease on imaging for at least 4 weeks prior to enrollment, discontinued systemic steroid therapy (≤10 mg/day prednisone or equivalent) for more than 4 weeks, and are asymptomatic, may be eligible; 12.Patients deemed by the investigator to be unable or unlikely to comply with the study protocol, restrictions, or requirements.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Estimated)
Dates: Start 2025-08-25 (Actual); Primary Completion 2026-12-30 (Estimated); Study Completion 2027-12-30 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival | Progression-free survival (PFS) analysis based on investigator assessment per RECIST 1.1, and will be assessed up to 2 years
  Progression free survival (PFS) refers to the time from recording the first chemotherapy treatment to the date of disease progression, as assessed by researchers.

SECONDARY OUTCOMES:
Overall Survival | The maximum time from receiving treatment to dying for any reason is 4 years.
  Overall survival (OS) refers to the time that researchers evaluate from recording the first chemotherapy to death (of any cause).
Objective response rate | Data obtained up until progression, or the last evaluable assessment in the absence of progression, will be assessed up to 1 years.
  Per Response Evaluation Criteria in Solid Tumors version 1.1 (RECIST 1.1) using Investigator assessments, is defined as the number (%) of patients with response of Complete Response or Partial Response, will be assessed up to 1 years.
Duration of Response | Duration of Response（DoR）analysis based on investigator assessment per RECIST 1.1, and will be assessed up to 1 years.
  Duration of Response（DoR）refers to the time from the first assessment as CR or PR to the first assessment as PD or (due to any reason) death.

CONTACTS AND LOCATIONS:
Locations (1):
- Tangdu Hospital Affiliated to the Fourth Military Medical University, Xi'an, Shannxi, China

IPD SHARING:
Plan to Share IPD: No